CLINICAL TRIAL: NCT01787942
Title: Investigating Abnormal Lipid Layer Thickness and Other Objective Dry Eye Parameters in Patients Seeking Blepharoplasty, and How They Change After Blepharoplasty
Brief Title: Investigating Abnormal Lipid Layer Thickness in Blepharoplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R974/83/2012; 2012/975/A (Other: Singhealth Centralised Institutional Review Board)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2013-02

CONDITIONS: Lipid Thickness
Keywords: Lipid thickness; Blepharoplasty; Tear break up time; Corneal staining

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blepharoplasty (Active Comparator): Participants under this group will undergo blepharoplasty from the oculoplastic clinic. These patients will form the "case" group of the cross-sectional study, and will be on follow-up for the prospective study.
  Interventions: Device: Tear Science LipiView
- Control (Placebo Comparator): Participants under this group will be recruited from the general ophthalmology clinic. These patients are cleared to have no lid disturbances in terms of function or anatomy, and will serve as the "control" group of the cross-sectional study.
  Interventions: Device: Tear Science LipiView

INTERVENTIONS:
Device: Tear Science LipiView — The LipiView is a non-invasive instrument that captures live, special and digital images of your tear film and measures its lipid content and quality. This is a standardized test that quantifies your lipid to help your eye doctor determine if you should undergo the LipiFlow procedure or other tear therapies that would treat your condition. In effect, the LipiView allows your eye doctor to visualize your tear films.

SUMMARY:
Deficiency in tear film lipid layer thickness (LLT) has been implicated in the development of dry eye symptoms, and is influenced to a significant degree by the anatomy and function of the eyelids. Patients who are considering blepharoplasty, even if it is for cosmetic reasons, may subtle differences in eyelid anatomy that pre-dispose them to having an abnormal tear lipid layer. Moreover, the changes in anatomy and contour of the eyelids following blepharoplasty introduce a whole new group of factors, such as an altered palpebral aperture and altered canthal fixation that can further change the eyelid's ability to maintain a healthy tear lipid layer, for better or for worse. Such changes in tear lipid layer can be detected with the aid of a newly acquired tear interferometer (LipiView, Tearscience Inc.), but has never been done in the context of blepharoplasty management. Due to the strong association between LLT and risk of dry eyes, we hope to investigate if there are significant differences in LLT and other objective dry eye parameters in two situations: 1) patients considering blepharoplasty as compared to other patients not considering such procedures 2) patients before and after undergoing blepharoplasty. The results of these investigations can go towards establishing LLT as an important objective parameter to account for before and after blepharoplasty.

DETAILED DESCRIPTION:
Study Objectives and Purpose

1. By cross-sectional analysis, determine if there are significant differences in average and SD of LLT in a group of patients who are considering blepharoplasty (cases) as compared to a group of patients from a general ophthalmology clinic who have no lid disturbances (controls).

2a. Via a prospective study, determine the average and standard deviation of LLT in a group of patients undergoing blepharoplasty, and how these change in a one month period after surgery.

2b. Identify, through the same prospective study, if factors such as age and gender are associated with the direction and magnitude of changes in LLT.

Study design:

Cross-sectional study and Prospective cohort study

Rationale:

1. A cross-sectional study comparing LLT, TBUT and corneal staining in patients who are about to undergo blepharoplasty against patients who have no complaints of any lid disturbances.
2. A prospective study observing changes in LLT, TBUT and corneal staining after blepharoplasty, and if age and gender was associated with these changes.

Methods:

30 patients who are about to undergo blepharoplasty will be recruited from the oculoplastic clinic. These patients will form the "case" group of the cross-sectional study, and will be on follow-up for the prospective study.

Another 30 patients will be recruited from the general ophthalmology (ECS) clinic. These patients are cleared to have no lid disturbances in terms of function or anatomy, and will serve as the "control" group of the cross-sectional study.

The following assessments will be performed for each patient who is recruited. For patients involved in the cross-sectional study, they will be assessed only once. For the patients involved in the prospective study, they will be assessed during the pre-surgery consultation, and at the standard post-surgery consultations at 1 week and 1 month after surgery

Procedures to be done

1. LLT measurement with LipiView tear interferometer
2. Fluorescein Dye Tear Break-up Time (TBUT)
3. Fluorescein Dye Corneal Staining

Duration of study: 1 year

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers that are medically fit and willing to participate in this study.
2. Volunteers who fit the criteria mentioned previously in the experimental design.

Exclusion Criteria:

1. Patients who are about to undergo cosmetic blepharoplasty.
2. Patients with other ocular surgeries pre-blepharoplasty that may have disturbed the ocular surface e.g. cataract phacoemulsification, pterygium removal.
3. Patients who experience major post-surgery side effects or complications unrelated to DES will be excluded from the study.
4. Patients with history of Parkinson's disease and other neurogenic conditions which interfere with blink rate.
5. Patients with proptosis or exophthalmos due to congenital reasons or Thyroid Eye Disease.
6. Patients who are on anti-histamine drugs.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Lipid layer thickness | 1 month
  Tear interferometry is non-invasive and is not unlike a standard slit-lamp examination of the eye. Patients will be asked to rest their chin on a chinrest and direct their sight at a single white-light source for 30 seconds. The same process will be repeated for another 30 seconds with the other eye. During this time, they are encouraged to blink at their comfortable pace. It is extremely safe and does not require contact of the ocular surface in any way.

SECONDARY OUTCOMES:
Tear break up time | 1 month
  Fluorescein dye is introduced onto the lower eyelid by a wetted fluorescein strip. The tear film will then be observed with blue light using a slit lamp to the point where it breaks. The time from the previous blink to the breaking of the tear film will be recorded to the nearest second.
Fluorescein Dye Corneal Staining | 1 month
  After fluorescein dye is introduced, the cornea will be examined for green stains indicating epithelial erosion, a sign of damage due to dryness. The number of green stains and their location on the cornea (superior, central, inferior, temporal, nasal fields) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, Phd, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre/ Singapore Eye Research Institute, Singapore, Singapore, Singapore